CLINICAL TRIAL: NCT03808415
Title: Jockey Club Tech-based Stroke Rehabilitation Programme - Hand of Hope
Brief Title: CUHK Jockey Club HOPE 4 Care Programme - Hand of Hope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor and Chairman, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018.399
Record Dates: First submitted 2018-12-20; First posted 2019-01-17 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMG-driven (Experimental): The hand training system functions as a biofeedback device which surface electromyography (EMG) sensors are used to capture the user's own muscle signals to activate the system for moving his/her paretic hand.
  Interventions: Device: EMG-driven

INTERVENTIONS:
Device: EMG-driven — The EMG signals are processed and can be visualized with visual feedback to make sure the user actively engaging throughout a therapy session.

SUMMARY:
The Hong Kong Jockey Club Charities Trust has supported CUHK to launch a three-year project 'CUHK Jockey Club HOPE4Care Programme' to implement four evidence-based advanced rehabilitation technologies in 40 local elderly day care centres and rehabilitation centres, to benefit the community.

The interactive intention-driven hand training robotic system is used for neuromuscular rehabilitation of the hand and forearm. This can help stroke survivors to regain their hand functions through motor relearning.

ELIGIBILITY:
Inclusion Criteria:

* at least six months after the onset of a unilateral ischemic brain injury or intracerebral haemorrhage
* upper-limb motor impairments due to stroke
* metacarpophalangeal and proximal interphalangeal joints of fingers can be extended to 180 degree passively
* spasticity during extension at the finger joints is lower than 3 as measured by the Modified Ashworth Scale
* detectable voluntary EMG signals from the flexor digitorum and extensor digitorum muscles of the paretic hand
* have sufficient cognition to follow the experimental instructions

Exclusion Criteria:

* have other neurological, neuromuscular, and orthopedic diseases
* have shoulder or arm contracture/pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | 3-month follow-up
Fugl-Meyer Assessment Upper Extremity (FMA-UE) | 3-month follow-up
Wolf Motor Function Test (WMFT) | 3-month follow-up

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu C, Ti CHE, Shi X, Yuan K, Leung TWH, Tong RK. Development and External Validation of a Motor Intention-Integrated Prediction Model for Upper Extremity Motor Recovery After Intention-Driven Robotic Hand Training for Chronic Stroke. Arch Phys Med Rehabil. 2025 Feb;106(2):206-215. doi: 10.1016/j.apmr.2024.08.015. Epub 2024 Aug 30. PMID 39218244